CLINICAL TRIAL: NCT06702618
Title: Evaluation of the Efficacy and Safety of TQB3616 Capsules Combined With Hormonal Therapy in a Phase II Clinical Trial for Cyclin-dependent Kinases 4 and 6（CDK4/6)Inhibitor-Resistant, Hormone Receptor(HR)-Positive, Human Epidermal Growth Factor Receptor 2(HER2)-Negative Recurrent/Metastatic Breast Cancer
Brief Title: Evaluation of TQB3616 Capsules in a Phase II Clinical Trial for Recurrent/Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-II-04
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3616 capsule+Fulvestrant Injection (Experimental)
  Interventions: Drug: TQB3616 capsule+Fulvestrant Injection

INTERVENTIONS:
Drug: TQB3616 capsule+Fulvestrant Injection — TQB3616 capsule is a CDK2/4/6 inhibitor and Fulvestrant injection is an anti-estrogen medication, and its pharmacological mechanism mainly exerts its therapeutic effect by inhibiting the action of aromatase.

SUMMARY:
Evaluation of the Efficacy and Safety of TQB3616 Capsules Combined with Hormonal Therapy in a Phase II Clinical Trial for Cyclin-dependent Kinases 4 and 6 (CDK4/6) Inhibitor-Resistant, HR-Positive, HER2-Negative Recurrent/Metastatic Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily join the study, sign the informed consent form, and have good compliance
* Aged 18 to 75 years, with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0~1; expected survival time of more than 3 months.
* Postmenopausal or premenopausal/perimenopausal female patients
* Progressed after prior treatment with CDK4/6 inhibitors
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Good major organ function
* Women of childbearing potential must agree to use contraception during the study and for 6 months after its completion.

Exclusion Criteria:

* Subjects with a previous pathological diagnosis of HER2-positive breast cancer.
* Subjects with inflammatory breast cancer or occult breast cancer.
* Subjects who have had or currently have other malignant tumors within 5 years prior to randomization.
* Subjects with unresolved toxicity (greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1) from prior treatment, excluding alopecia.
* Subjects who have undergone major surgical procedures, incisional biopsies, or significant traumatic injuries within 28 days prior to the first dose.
* Subjects with non-tumor-related unresolved wounds, ulcers, or fractures.
* Subjects with multiple factors affecting oral medication intake and absorption.
* Subjects with arterial or deep vein thrombotic events within 6 months prior to the first dose.
* Subjects with ≥ Grade 2 myocardial ischemia or myocardial infarction, arrhythmia, angina requiring anti-anginal medication, clinically significant valvular heart disease, or uncontrolled hypertension.
* Subjects with a history of interstitial lung disease/pneumonitis (non-infectious) requiring steroid intervention or currently having interstitial lung disease/pneumonitis, or subjects with suspected interstitial lung disease/pneumonitis on screening imaging that cannot be excluded.
* Subjects with active or uncontrolled serious infections (≥CTCAE Grade 2 infection) or unexplained fever >38.5°C within 28 days prior to the first dose.
* Subjects with a history of abuse of psychotropic drugs that cannot be abstained from or those with psychiatric disorders.
* Subjects with (pseudo) cirrhosis, active hepatitis.
* Subjects with renal failure requiring hemodialysis or peritoneal dialysis.
* Subjects with a history of immunodeficiency diseases, organ transplants, or hematopoietic stem cell transplants.
* Subjects who have previously received fulvestrant or other oral Selective Estrogen Receptor Degrader (SERD) class drugs.
* Subjects who have previously received anti-HER2 therapy.
* Subjects who have previously received antibody-drug conjugate therapy.
* Subjects who have participated in other anti-tumor clinical trials and taken investigational drugs within 4 weeks prior to the first dose.
* Subjects judged by the investigator to have serious accompanying diseases that severely endanger the safety of the subject or affect the completion of the study, or subjects who are deemed unsuitable for enrollment for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Baseline up to 12 months
  The proportion of patients achieving complete response and partial response among the total evaluable cases.

SECONDARY OUTCOMES:
Progression Free Survival | Baseline up to 12 months
  Progression Free Survival (PFS) is defined as the length of time from the start of treatment until the disease progresses or the patient dies from any cause.
Duration of Response | Baseline up to 12 months
  The time from the first assessment of the tumor as a complete response or partial response to the first occurrence of disease progression or death from any cause.
Disease Control Rate | Baseline up to 12 months
  The percentage of subjects with a complete response, partial response, or stable disease as determined by RECIST 1.1.
Clinical Benefit Rate | From the first dose to complete response, partial response, or stable disease for ≥24 weeks
  The percentage of subjects with a complete response, partial response, or stable disease for ≥24 weeks as determined by RECIST 1.1.
Overall Survival | Baseline up to 24 months
  The time from the start of initial treatment to death from any cause
Adverse event (AE) | From the subject's signing of the informed consent form to 28 days after the last dose or the start of new anti-tumor therapy (whichever occurs first)
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - The First Affilliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hostipal, Harbin, Heilongjiang
  - Luohe Central Hospital, Luohe, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Hai'an People's Hospital, Nantong, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Cancer Hospital of Shandong First Medical University(Shandong Cancer Institute, Shandong Cancer Hospital), Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality